CLINICAL TRIAL: NCT00230750
Title: A Randomized, Double-Blinded, Placebo-Controlled Phase I/II, Dose-Ranging Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Healthy Elderly Adults
Brief Title: Inactivated Influenza A/H5N1 Vaccine in the Elderly
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-076
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2008-09

CONDITIONS: Influenza
Keywords: influenza, elderly, vaccine, H5N1, parent protocol
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 2 (Experimental): 100 subjects to receive 90 mcg of inactivated influenza A/H5N1 vaccine on days 0, 28, and 6 months following the 1st vaccination.
  Interventions: Biological: Influenza A/H5N1 Vaccine
- 3 (Placebo Comparator): 40 subjects to receive saline placebo on days 0, 28, and 6 months following the 1st vaccination.
  Interventions: Drug: Placebo
- 1 (Experimental): 100 subjects to receive 45 mcg of inactivated influenza A/H5N1 vaccine on days 0, 28, and 6 months following the 1st vaccination.
  Interventions: Biological: Influenza A/H5N1 Vaccine

INTERVENTIONS:
Biological: Influenza A/H5N1 Vaccine — Monovalent subvirion H5N1 vaccine (HA of A/Vietnam/1203/04) provided in unit-dose vials containing 90-mcg/mL. Dosages: 45 mcg or 90 mcg administered intramuscularly.
  Arms: 1; 2
Drug: Placebo — Saline placebo.
  Arms: 3

SUMMARY:
The purpose of this research study is to compare how the body reacts to different strengths of a new H5N1 flu vaccine. Researchers will also look at how antibodies are made after subjects receive the H5N1 flu vaccine. Participants will include at least 240 healthy males and females, aged 65 and older. The vaccine is given as an injection or shot in the arm. Subjects will receive 3 doses of vaccine at Day 0, Month 1 and Month 6. There are 2 different doses of the new H5N1 vaccine that will be given in this study. There is also a chance that a subject may receive a placebo (dummy) injection of saltwater instead of the flu vaccine. Study procedures will include physical exams and blood sample collections. Additionally, participants will complete a memory aid card to document daily temperatures and any symptoms experienced for a week after receiving vaccine. The length of participation in this study will be approximately 14 months.

DETAILED DESCRIPTION:
The goals of this study are to compare the safety, reactogenicity, and immunogenicity of two dose levels of monovalent subvirion influenza A/H5N1 virus vaccine administered by injection to healthy elderly adults aged 65 years and older. Researchers hypothesize that a dose of either 45 micrograms or 90 micrograms of H5N1 vaccine will be well tolerated and result in acceptable immunogenicity. Thus, the primary goal of this study is to determine the lowest dose level of H5N1 that will result in an acceptable proportion of subjects achieving a potentially protective postvaccination antibody titer combined with an acceptable safety profile. The study will enroll at least 240 (and up to 260) healthy ambulatory male and female subjects aged 65 and older, in the United States, may be enrolled. Three doses of the vaccine at 2 dose levels (45 micrograms or 90 micrograms) or saline placebo will be administered 28 days apart for the first two doses. The third dose will be given six months after the first dose. Serum hemagglutination inhibition (HAI) and neutralizing antibody titers will be assessed approximately 1 month after receipt of each dose and 6 month after first and third doses. The primary objectives of the study are: to determine the dose-related safety of intramuscular (IM) subvirion inactivated H5N1 vaccine in healthy elderly adults (65 years of age and older); to determine the immunogenicity of IM subvirion inactivated H5N1 vaccine approximately 1 month following receipt of 2 doses of vaccine; and to provide information for the selection of the best dose level(s) for further studies. The secondary objective is to determine the immunogenicity of IM subvirion inactivated H5N1 vaccine approximately 1 and 6 months following receipt of first and third doses of the vaccine. The primary endpoints include: adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessments); proportion of subjects achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus 28 days after receipt of second dose of vaccine (approximately Day 56); geometric mean titer (GMT) and the frequency of 4-fold or greater increases in neutralizing antibody titers 28 days after receipt of second dose of vaccine (approximately Day 56). The secondary endpoints include: development of serum antibody responses against antigenically drifted variants of H5N1 influenza virus and geometric mean titer and the frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) and neutralizing antibody titer 1 and 6 months after receipt of first and third dose of vaccine. The duration of the study will be approximately 15 months (approximately 14 months for each subject). This study is linked to DMID protocols 07-0022 and 05-0006.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adult aged 65 and older.
* Is in good health, as determined by vital signs (heart rate <100 bpm, blood pressure [systolic less than or equal to 160 mm Hg and diastolic less than or equal to 90 mm Hg] oral temperature < 100 degrees F), medical history to ensure stable medical condition, and a targeted physical examination based on medical history.
* Able to understand and comply with planned study procedures.
* Provides informed consent prior to any study procedures and is available for all study visits.

Exclusion Criteria:

* Has a known allergy to eggs or other components of the vaccine or sensitivity to latex.
* Is undergoing immunosuppression as a result of an underlying illness or treatment.
* Has any malignancy (excluding nonmelanotic skin cancer) or lymphoproliferative disorder diagnosed or treated actively during the past 5 years.
* Is using oral or parenteral steroids, high-dose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Has a history of alcohol abuse or drug abuse (including chronic pain medication) in the last 5 years.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include, but are not limited to: history of significant renal impairment (dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease); subjects with diabetes mellitus, well-controlled with oral agents may enroll as long as there has been no dose adjustment within the past 6 months; insulin-dependent diabetes is excluded; cardiac insufficiency, if heart failure is present (New York Heart Association Functional Class III or IV); arteriosclerotic event during the 6 months prior to enrollment (e.g., history of myocardial infarction, stroke, recanalization of femoral arteries, or transient ischemic attack).
* Has a history of severe reactions following immunization with influenza virus vaccines.
* Has an acute illness, including an oral temperature greater than 100.0 degrees F, within 1 week prior to vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the 14-month study period.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Has any diagnosis of dementia or associated concomitant medications (e.g., Aricept) used for treating dementia.
* Has known Latex allergy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 261 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) and the frequency of 4-fold or greater increases in neutralizing antibody titers 28 days after receipt of second dose of vaccine. | Approximately day 56.
Proportion of subjects achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus 28 days after receipt of second dose of vaccine. | Approximately day 56.
Adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessments). | Adverse events will be collected for 28 days following each dose of vaccine. Serious adverse events will be collected throughout the study through month 13.

SECONDARY OUTCOMES:
Development of serum antibody responses against antigenically drifted variants of H5N1 influenza virus. | Blood samples for serum assays will be collected at day 0 and at days 28, 56, month 6, 7 and 13 after the first immunization.
Geometric mean titer and the frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) and neutralizing antibody titer 1 and 6 months after receipt of first and third dose of vaccine. | Blood samples for serum assays will be collected at day 0 and at days 28, 56, month 6, 7 and 13 after the first immunization.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Center For Vaccine Research, Torrance, California
  - University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee